CLINICAL TRIAL: NCT04129840
Title: Identifying Most Effective Treatment Strategies to Control Arterial Hypertension in Sub-Saharan Africa - A Randomized Controlled Trial
Brief Title: Identifying Most Effective Treatment Strategies to Control Arterial Hypertension in Sub-Saharan Africa
Acronym: coArtHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Fund for Scientific Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-00817; qu19Weisser
Record Dates: First submitted 2019-10-03; First posted 2019-10-17 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Arterial Hypertension
Keywords: antihypertensive treatment
MeSH Terms: conditions — Hypertension | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The intervention is a treatment algorithm (comparing two combination treatment strategies with the World Health Organization (WHO) standard and not an individual drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1: dual combination (Active Comparator): dual combination of half-dose Calcium Channel Blocker (CCB) and Angiotensin II Receptor Blocker (ARB), dosage increases at 4 and 8 weeks if target blood pressure is not reached at the respective time point
  Interventions: Other: dual combination
- Intervention 2: triple combination (Active Comparator): triple combination of quarter-dose of Calcium Channel Blocker (CCB), Thiazide diuretic (TZD) and Angiotensin II Receptor Blocker (ARB) with dosage increases of all drugs at 4 and 8 weeks, if target blood pressure is not reached at the respective time point
  Interventions: Other: triple combination
- Standard of care (Placebo Comparator): start normal dose Calcium Channel Blocker (CCB), add Thiazide diuretic (TZD) after 4weeks and increase of TZD dosage after 8 weeks, if target blood pressure is not reached at the respective time point
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: dual combination — Participants will be started on a dual therapy with half dose of CCB and an ARB. If needed, a) the dose of the CCB will be increased at 4 weeks, and b) the dose of the ARB at 8 weeks, if blood pressure remains uncontrolled ((if target blood pressure is not achieved at this time point (target blood pressure defined as clinic BP </=130/80mmHg in patients <65years and </=140/90mmHg in patients >65years)
  Arms: Intervention 1: dual combination
Other: triple combination — Participants will be started with low dose (1/4) triple combination treatment with CCB, TZD and ARB. If uncontrolled after 4 weeks, dosages of all drugs will be doubled. If after 8 weeks still uncontrolled dosage will be increased to full dose of all three drugs ((if target blood pressure is not achieved at this time point (target blood pressure defined as clinic BP </=130/80mmHg in patients <65years and </=140/90mmHg in patients >65years)
  Arms: Intervention 2: triple combination
Other: Standard of care — Participants will be started on regular dose of CCB with a) addition of TZD at 4 weeks, if needed, b) increase of dose of TZD after 8 weeks, if needed (if target blood pressure is not achieved at this time point (target blood pressure defined as clinic BP </=130/80mmHg in patients <65years and </=140/90mmHg in patients >65years)
  Arms: Standard of care

SUMMARY:
This study is to compare the effectiveness of three different antihypertensive treatment strategies for reaching a target blood pressure (clinic BP) of </= 130/80 mmHg among patients <65years of age and </= 140/90 mmHg among patients >/=65years of Age in HIV-positive and HIV-negative patients with uncomplicated arterial hypertension in rural Tanzania and Lesotho.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive and negative patients of African descent and black ethnicity with a documented uncomplicated, untreated arterial hypertension (blood pressure >/=140/90 mmHg) diagnosed at one of the 2 study sites

Exclusion Criteria:

* Current hospitalization for any reason
* Not of African descent
* Refusal of an HIV-test or indeterminate HIV test result
* History of cardiovascular event in the last month (anginal pain, stroke, myocardial infarction or diagnosis by a doctor)
* Symptomatic arterial hypertension (blood pressure >/=180/110 mmHg plus headache or chest pain) or acute cardiovascular event
* acute disease, (e.g. fever >37.5°C or other signs of acute concomitant infection; Dyspnea/respiratory distress; Acute pain)
* Clinical signs of hypertension-mediated organ damage (heart failure, bilateral pitting edema, bilateral crackles or pleural effusion, distended jugular veins, ischemic heart disease (anginal pain on exertion), signs of current ischemic/hemorrhagic stroke (hemiparesis, loss of consciousness)
* Pregnancy (test required for females 18-45years of age)
* Non-consenting or inability to come for follow-up visits
* creatinine clearance </=30ml/min by Chronic Kidney Disease Epidemiology Formula (CK-EPI) estimation and measurement with a point-of care creatinine from capillary blood

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1268 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reaching a target blood pressure | at 12 weeks after enrolment
  Proportion of patients reaching a target blood pressure (clinic blood pressure) of </=130/80 mmHg in patients <65years of age and </=140/90 mmHg in patients >65years of age

SECONDARY OUTCOMES:
Proportion of patients reaching a target blood pressure | at 4, 8 and 24 weeks after enrolment
  Proportion of patients reaching a target blood pressure (clinic blood pressure) of </=130/80mmHg in patients <65years of age and </=140/90mmHg in patients >65years of age
Change in blood pressure (mmHg) | at 4, 8, 12, 24 weeks after enrolment
  Change in blood pressure (change from enrolment) (mmHg)
Proportion of patients with treatment adaptations made to the primary treatment | within 12 weeks after enrolment
  Proportion of patients with treatment adaptations made to the primary treatment (dose increases and/or drug additions)
Number of treatment adaptations per patient made to the primary treatment | within 12 weeks after enrolment
  Number of treatment adaptations per patient made to the primary treatment
Time until first target blood pressure of </=130/80 mmHg in patients <65years of age and </=140/90mmHg in patients >65years of age | within 24 weeks after enrolment
  Time until first target blood pressure of </=130/80 mmHg in patients <65years of age and </=140/90mmHg in patients >65years of age
Proportion of patients with major cardiovascular endpoints | within 24 weeks after enrolment
  Proportion of patients with major cardiovascular endpoints such as death, stroke, myocardial infarction, heart failure)
Proportion of patients with changes in surrogate markers for hypertension-mediated organ damage | within 24 weeks after enrolment
  Proportion of patients with changes in surrogate markers for hypertension-mediated organ damage (resolving, newly occurring or worsening)
Proportion of patients lost to follow up or stopped treatment | within 24 weeks after enrolment
  Proportion of patients lost to follow up or stopped treatment
Proportion of patients with at least one grade 3/4 adverse event | within 24 weeks after enrolment
  Proportion of patients with at least one grade 3/4 adverse event
Proportion of patients with at least one severe adverse event | within 24 weeks after enrolment
  Proportion of patients with at least one severe adverse event
Proportion of patients who were non-adherent to drugs | at 12 weeks after enrolment
  Proportion of patients who were non-adherent to drugs (<90% pill count or <90% of self-reported drug intake)
Reasons for non-adherence assessed by pill count (descriptive analysis) | within 24 weeks after enrolment
  Reasons for non-adherence assessed by pill count (descriptive analysis)
Cost-effectiveness of the 3 treatment algorithms | within 24 weeks after enrolment
  Cost-effectiveness of the 3 treatment algorithms
Proportion of patients with white coat hypertension, as determined by 24h ambulatory blood pressure measurement | within 12 weeks after enrolment
  Proportion of patients with white coat hypertension, as determined by 24h ambulatory blood pressure measurement
Proportion of patients with blood pressure control determined by 24h ambulatory blood pressure measurement (24h mean blood pressure <130/80mmHg irrespective of age) | within 12 weeks after enrolment
  Proportion of patients with blood pressure control determined by 24h ambulatory blood pressure measurement (24h mean blood pressure <130/80mmHg irrespective of age)
Reasons for non-adherence assessed by self-report (descriptive analysis) | within 24 weeks after enrolment
  Reasons for non-adherence assessed by self-report (descriptive analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Maja Weisser Rohacek, PD Dr., Principal Investigator — Division of Infectious Diseases & Hospital Epidemiology, University Hospital Basel
Locations (3):
- SolidarMed Lesotho, Mokhotlong Government Hospital, Mokhotlong, Lesotho
- Division of Infectious Diseases & Hospital Epidemiology; University Hospital Basel, Basel, Switzerland
- St. Francis Referral Hospital/ Ifakara Health Institute, Ifakara, Morogoro, Tanzania

REFERENCES:
- [Derived] Mapesi H, Rohacek M, Vanobberghen F, Gupta R, Wilson HI, Lukau B, Amstutz A, Lyimo A, Muhairwe J, Senkoro E, Byakuzana T, Nkouabi J, Mbunda G, Siru J, Tarr A, Ramapepe E, Mphunyane M, Oehri J, Nemtsova V, Yan X, Bresser M, Glass TR, Paris DH, Fink G, Gingo W, Labhardt ND, Burkard T, Weisser M. Treatment Strategies to Control Blood Pressure in People With Hypertension in Tanzania and Lesotho: A Randomized Clinical Trial. JAMA Cardiol. 2025 Apr 1;10(4):321-333. doi: 10.1001/jamacardio.2024.5124. PMID 39878989
- [Derived] Mapesi H, Gupta R, Wilson HI, Lukau B, Amstutz A, Lyimo A, Muhairwe J, Senkoro E, Byakuzana T, Mphunyane M, Bresser M, Glass TR, Lambiris M, Fink G, Gingo W, Battegay M, Paris DH, Rohacek M, Vanobberghen F, Labhardt ND, Burkard T, Weisser M. The coArtHA trial-identifying the most effective treatment strategies to control arterial hypertension in sub-Saharan Africa: study protocol for a randomized controlled trial. Trials. 2021 Jan 21;22(1):77. doi: 10.1186/s13063-021-05023-z. PMID 33478567